CLINICAL TRIAL: NCT00013416
Title: Measurement and Prediction of Outcomes of Amplification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2002R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Hearing Impaired
Keywords: Hearing loss, hearing aid, amplification
MeSH Terms: conditions — Hearing Loss | interventions — Hearing

INTERVENTIONS:
Procedure: Hearing

SUMMARY:
The long-term goal of this research program is to develop methods to predict both the benefit and the satisfaction that hearing-impaired patients will derive from auditory amplification in daily life. This proposal has three primary objectives: (1) To determine the influence of extra-audiological variables, such as personality attributes and expectations, on the subjective outcomes of hearing aid fittings, (2) To establish a scientific basis for selection, administration, and interpretation of self-report measures of hearing aid fitting outcome, (3) To resolve the long-standing debate about the efficacy of using clinically measured loudness perception data in hearing aid prescriptions.

DETAILED DESCRIPTION:
The long-term goal of this research program is to develop methods where by clinicians can predict both the benefit and the satisfaction that individual hearing-impaired patients will derive from amplification in daily life. The present proposal continues the research directions pursued in several cycles of previous RR&D funding from 1986 to 1996. This proposal has three primary objectives: (1) To determine the influence of extra-audiological variables, such as personality attributes and expectations, on the subjective outcomes of hearing aid fittings, (2) To establish a scientific basis for selection, administration, and interpretation of self-report measures of hearing aid fitting outcome, (3) To resolve the long-standing debate about the efficacy of using clinically measured loudness perception data in hearing aid prescriptions.

HYPOTHESES:

1. Inter-subject differences in personality traits, coping style, and/or expectations account for a significant and substantial amount of the variance in hearing aid fitting outcomes, independent of hearing impairment and fitting strategy.
2. Prediction of hearing aid fitting outcomes will be substantially improved if the prediction model includes extra-audiological data as well as data on impairment and hearing aid.
3. The post-fitting time course of hearing aid fitting outcome data is different for different outcome variables.
4. Self-report hearing aid fitting outcomes are stable after 3 months of hearing aid use.
5. Fitting outcomes are optimized for individuals with unpredictable loudness perception when clinically measured loudness data are used in the hearing aid fitting protocol.

PROCEDURES: Investigations will explore:(1)the determinants and characteristics of subjective outcome variables, and (2) the value of individual loudness data in hearing aid fitting. Subjects will be elderly men and women with bilateral sensorineural hearing loss. The work will be performed at the Memphis VAMC Hearing Aid Research Laboratory.

Determinants and characteristics of subjective outcome variables. When self-reports are used to evaluate hearing aid fitting outcome, it is assumed that the data primarily reflect the efficacy of the hearing aid and the fitting strategy. There is a lack of information about the extent to which other variables might impact self-report data. We will explore this topic with 120 potential hearing aid wearers, followed from their initial expression of interest in amplification through the entire fitting process and for six months after the fitting. Data describing a range of pre-fitting variables as well as hearing impairment, and hearing aid fitting will be collected in a consortium of six clinical sites (including 5 VA sites) coordinated from the Memphis laboratory. The Memphis research team will complete data collection with each subject by collecting outcome data at three post-fitting intervals.

ELIGIBILITY:
Hearing-impaired patients

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 1999-10; Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D., Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), rehabilitation Research & Development Service; Nancy Rocheleau, Program Analyst — Department of Veterans Affairs, Program Analysis and Rreview Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Memphis, Memphis, Tennessee, United States